CLINICAL TRIAL: NCT05067530
Title: Cyclin dEpendent Kinase in tRiple nEGatIVe brEast canceR - a "Window of Opportunity" Study
Acronym: CAREGIVER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBK 171/1/2021; 2021-001556-33 (EudraCT Number)
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Triple Negative Breast Neoplasms
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — palbociclib; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, multicenter, open, five-arm study with unequal allocation ratios of 1:1:2:1:2 (palbociclib : paclitaxel : palbociclib + paclitaxel : carboplatin : carboplatin + paclitaxel)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CDK4/6 inhibitor alone: Palbociclib (IMP) (Experimental): Palbociclib alone (125 mg orally (PO) per day, days 1-14)
  Interventions: Drug: Palbociclib
- Chemotherapy alone: Paclitaxel (Active Comparator): Paclitaxel alone (80 mg/m^2 intravenously (IV), day 1, 8, 15 and 22)
  Interventions: Drug: Paclitaxel
- CDK4/6 inhibitor + chemotherapy: Paclitaxel + Palbociclib (Experimental): Paclitaxel (80 mg/m^2 IV, day 1, 8, 15 and 22) + Palbociclib (125 mg PO per day, days 1-21)
  Interventions: Drug: Palbociclib; Drug: Paclitaxel
- Chemotherapy alone: Carboplatin (Active Comparator): Carboplatin alone (area under the curve (AUC) 2 IV, day 1, 8, 15 and 22)
  Interventions: Drug: Carboplatin
- CDK4/6 inhibitor + chemotherapy: Carboplatin + Palbociclib (Experimental): Carboplatin (AUC 2 IV, day 1, 8, 15 and 22) + Palbociclib (125 mg PO per day, days 1-21)
  Interventions: Drug: Palbociclib; Drug: Carboplatin

INTERVENTIONS:
Drug: Palbociclib — CDK4/6 inhibitor
  Other Names: Ibrance
  Arms: CDK4/6 inhibitor + chemotherapy: Carboplatin + Palbociclib; CDK4/6 inhibitor + chemotherapy: Paclitaxel + Palbociclib; CDK4/6 inhibitor alone: Palbociclib (IMP)
Drug: Paclitaxel — Chemotherapy
  Arms: CDK4/6 inhibitor + chemotherapy: Paclitaxel + Palbociclib; Chemotherapy alone: Paclitaxel
Drug: Carboplatin — Chemotherapy
  Arms: CDK4/6 inhibitor + chemotherapy: Carboplatin + Palbociclib; Chemotherapy alone: Carboplatin

SUMMARY:
CAREGIVER is a prospective, randomized, multicenter, open, five-arm study with unequal allocation ratios of 1:1:2:1:2 (palbociclib : paclitaxel : palbociclib + paclitaxel : carboplatin : carboplatin + paclitaxel). Study will be performed in untreated patients with triple-negative breast cancer (TNBC). Potential candidates without previously established diagnosis of TNBC will be included in a Pre-screening Phase, when a biopsy of breast tumor will be taken to confirm the diagnosis of cancer, select patients with TNBC and collect tissue for translational research.

ELIGIBILITY:
Inclusion Criteria:

* females or males >18 years old at the time of informed consent signature;
* diagnosis of potentially resectable or de novo metastatic (stage II-IV) invasive carcinoma of the breast;
* eligible for standard neoadjuvant or palliative paclitaxel and/or carboplatin-based chemotherapy as determined by Investigator;
* triple negative tumor defined as:

  * hormone receptor-negative (<1% ER/PgR expression);
  * HER2-negative (Immunohistochemistry (IHC) score ≤1 or IHC score =2 and negative for the amplification by in situ hybridization);
* multicentric/multifocal disease is allowed, provided that all lesions have been biopsied and their phenotype has been confirmed pathologically as TNBC;
* no previous anticancer therapy for this malignancy;
* clinically or radiographically measurable disease (discrete lesion only, enhancement is not included) within the breast, that can be biopsied, defined as longest diameter >2 cm;
* multicentric or multifocal disease is allowed if at least 1 lesion is >2 cm;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* adequate bone marrow and organ function as defined by the following local laboratory values:
* hemoglobin ≥9 g/dL;
* absolute neutrophil count (ANC) ≥1500/μL;
* platelets ≥100,000/μL;
* total bilirubin ≤ institutional upper limit of normal (ULN), unless diagnosis of Gilbert syndrome;
* aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5x ULN;
* creatinine ≤ ULN OR creatinine clearance ≥50 mL/min per Cockcroft-Gault equation for patients with creatinine levels greater than ULN.
* blood glucose level <120 mg/dL after at least 6 hours of fasting;
* standard 12-lead electrocardiogram (ECG) without clinically significant abnormalities;
* ability to undergo contrast-enhanced MRI;
* ability to swallow and retain oral medication;
* all study participants of child-bearing potential must agree to use adequate contraceptive methods prior to study entry, during the study and for the following 3 weeks (females) or 14 weeks (males);
* prior chemotherapy, other targeted anticancer therapies, or prior radiation therapy (outside of treated breast) for other malignancy treated with radical intent is allowed, provided the treatment was completed ≥1 year before informed consent signature;
* prior bisphosphonate therapy is allowed;
* willing and able to undergo all the procedures required by the study protocol;
* provision of written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* inflammatory breast cancer;
* prior systemic treatment for this malignancy;
* prior treatment with CDK4/6 inhibitor;
* known hypersensitivity to study medications or any of their excipients;
* major surgery or radiotherapy (apart from limited field radiotherapy for symptom control) within 14 days prior to randomization;
* concurrent invasive malignancy;
* known HIV, active HBV or HCV infection;
* active autoimmune disease requiring ongoing immunosuppressive therapy;
* history of allotransplantation;
* concurrent treatment with systemic immunosuppressive agents, including steroids, within 3 weeks of enrolment;
* presence of implants or devices not compatible with MRI;
* pregnant or nursing female participants;
* receiving strong inhibitors or inducers of CYP3A4/5 or medications with narrow therapeutic window that are predominantly metabolized through CYP3A4/5;
* impairment of GI function that may significantly alter the absorption of the oral trial treatments;
* unwilling or unable to follow protocol requirements, including obligatory biopsies;
* any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drugs;
* any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment, contraindicate patient participation in the clinical trial or compromise compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
Early metabolic response | Day 27 (± 3 days)
  Difference in early (i.e., after three weeks of therapy, 1 cycle) metabolic response to treatment in chemotherapy-containing arms (chemotherapy ± palbociclib), as assessed by Blinded Central Review comparison of decrease in SUVmax between baseline and Day 27 (± 3 days) 18-fluoro-2-deoxy-d-glucose (18FDG) positron emission tomography - computed tomography (PET-CT). Primary analysis will include comparison between chemotherapy + palbociclib vs chemotherapy alone arms.

SECONDARY OUTCOMES:
SUVmax change | Day 27 (± 3 days)
  Difference in proportion of patients with SUVmax change above the predefined cut-off of 30% between chemotherapy + palbociclib vs chemotherapy alone arms.
Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) | Day 27 (± 3 days)
  Difference in Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST)-based peak standardized uptake value corrected for lean body mass in a spherical 1 cm3 volume of interest (SULpeak) decrease in PET-CT between chemotherapy + palbociclib vs chemotherapy alone arms.
Metabolic tumor volume (MTV) difference | Day 27 (± 3 days)
  Difference in metabolic tumor volume (MTV) regression between chemotherapy + palbociclib vs chemotherapy alone arms.
Tumor diameter change | Day 27 (± 3 days)
  Maximum tumor diameter change in largest continuous tumor mass based on MR imaging.
Change in tumor characteristic | Day 27 (± 3 days)
  Change in tumor characteristic in Day 27 biopsy (presence of viable cancer cells).
Treatment toxicity | Day 27 (± 3 days)
  Treatment toxicity (with special attention to myeloid toxicity to explore potential myeloprotective activity): number and severity of adverse events (AEs); toxicity will be described according to ICD-10 codes and graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).

CONTACTS AND LOCATIONS:
Locations (6):
- Poland (6):
  - Wielkopolskie Centrum Onkologii im. Marii Skłodowskiej-Curie, Oddział Onkologii Klinicznej i Immunoonkologii z Pododdziałem Dziennym, Poznan, Greater Poland Voivodeship
  - Dolnośląskie Centrum Onkologii we Wrocławiu, Oddział Onkologii Klinicznej/Chemioterapii, Poradnia Chemioterapii; Leczenie Nowotworów Piersi, Wroclaw, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie, Warsaw, Masovian Voivodeship
  - SP ZOZ Opolskie Centrum Onkologii im. Prof. Tadeusza Koszarowskiego, Opole, Opole Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie, Państwowy Instytut Badawczy, Oddział w Gliwicach, Gliwice, Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No